CLINICAL TRIAL: NCT06269653
Title: Measuring Protein Turnover in Humans Across the Lifespan by Metabolic Labeling With Deuterium Oxide
Status: Recruiting | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001944; 001944-AG
Record Dates: First submitted 2024-02-16; First posted 2024-02-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12-12

CONDITIONS: Healthy Volunteers
Keywords: PROTEIN TURNOVER; Metabolic; Mononucleated Cells; Mitochondrial; Peripheral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Healthy Individuals: 20 - 29 years of age: Age group: 20 -29 (3 men and 3 women)
- Healthy Individuals: 30 - 39 year of age: Age group: 30 - 39 (3 men and 3 women)
- Healthy Individuals: 40 - 49 years of age: Age group 40 - 49 (3 men and 3 women)
- Healthy Individuals: 50 - 59 years of age: Age group: 50 - 59 (3 men and 3 women)
- Healthy Individuals: 60 - 69 years of age: Age group: 60 - 69 (3 men and 3 women)
- Healthy Individuals: 70 +: Age group: 70+ (3 men and 3 women)

SUMMARY:
Background:

Proteins are essential to the health and structure of the cells that make up body tissues. Most proteins become damaged over time and are replaced with new ones. This process is called "protein turnover." Stress, disease, and aging can affect this process. Researchers want to better understand how aging affects protein turnover.

Objective:

To measure rates of protein turnover in healthy adults.

Eligibility:

Healthy people aged 20 years and older with a body mass index between 20 and 30.

Design:

Participants will have 6 study visits over 4 to 6 weeks. They will fast 12 hours before each visit.

Participants will be screened. They will have a physical exam, with blood and urine tests and tests of their heart function. They will lie down while blood pressure cuffs are used on their arms and legs.

Participants will be given bottles of heavy water to drink at home on a schedule for 21 days. Each bottle holds about 3.5 tablespoons. Heavy water is odorless, colorless, and tasteless, like normal drinking water. It is safe to drink and has been used in research for many years.

Participants will have tests during study visits, including:

Imaging scans of a leg.

Exercise on a treadmill.

Biopsies of muscle, skin, and fat: Small samples of tissue will be cut from the calf and abdomen.

Resting metabolic rate: Participants will lie still and breathe into a mask for 20 minutes.

Knee/grip strength: Participants will do strength tests with their legs. They will squeeze a device with their hands.

D3-Creatine: Participants will take 1 pill of D3-Creatine, which occurs naturally in muscle.

DETAILED DESCRIPTION:
Study Description:

A sophisticated biological system of quality control ensures that proteins are maintained in all cells in the right absolute and relative quantities and their architectural characteristics are preserved so that they can perform their biological function. There is evidence from animal models that the half-life of a subset of proteins is longer with aging so that aggregated proteins are retained for longer time than in younger individuals, leading to reduced cellular function. On the other hand, other proteins such as mitochondrial proteins are damaged at a higher rate and are expected to turnover faster to maintain function. This study is aimed at evaluating the half-life of a range of proteins in muscle, peripheral blood mononucleated cells (PBMCs), and skin in participants of different ages and tests the hypothesis that for specific proteins, older persons have different protein turnover than younger persons and that the effect of aging on proteins half-life is also dependent on the specific tissue considered.

Objectives:

Primary Objective: To measure the turnover proteins in humans across tissues, age, and sex.

Secondary Objective: To test the hypothesis that older age is associated with diminished protein turnover.

Endpoints:

Primary Endpoint: The primary endpoint of this study is to characterize the turnover of different proteins in human skeletal muscle.

Secondary Endpoint: The secondary endpoint of this study is to assess whether the turnover of proteins in skeletal muscle is significantly associated with aging.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, age >= 20years.
* BMI >20 and <30.
* In good general health as evidenced by medical history/exam/laboratory.
* IL6< 3.5 pg/mL.
* Ankle Brachial Index (ABI) > 0.9.
* No history of increased bleeding due to either a known medical condition or an undiagnosed cause.
* Does not currently smoke/tobacco use.
* Eligible for muscle biopsy procedures.
* Is not allergic to lidocaine or other local anesthetics.
* Able to speak and read English.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Routinely taking (more than 2x/week) non-steroidal anti-inflammatory agents (NSAIDs) and unwilling to stop taking them for the duration of the study.
* Taking medications that could increase the chance of bleeding such as anticoagulants/antiplatelet such as Coumadin, Plavix, and Heparin. Low dose (81mg) aspirin use is okay.
* Is unable to reach down to perform wound care of the lower legs.
* Has laboratory evidence of diabetes at screening (fasting glucose >= 126) and/or diabetes requiring treatment, or treatment with any glucose lowering drug(s).
* Has current or history of inflammatory and/or autoimmune diseases.
* History of keloid formation.
* Researchers are unable to access biopsy sites due to conditions such as wounds, rashes, or large deposits of adipose tissue.
* Is on treatment with an investigational drug or other intervention within 8 weeks of enrollment.
* Has any chronic disease that the study PI considers as a significant comorbidity that affects health and life expectancy.
* Has established genetic diseases such as sickle cell, hemochromatosis (iron overload), cystic fibrosis or Ehlers-Danlos syndrome (connective tissue disorder).
* Has autoimmune diseases such as Hashimoto s thyroiditis, Myasthenia Gravis, or Rheumatoid arthritis.
* Has severe mobility disability as evidenced by inability to walk without aids, perform activities of daily living and to reach down to lower legs to perform wound care.
* Has had active cancer on treatment in the last 10 years.
* Has muscle-skeletal conditions due to diseases or traumas (that cause pathological weakness and/or chronic pain).
* Has any medical condition that requires absolute and continuous need for long term treatment with antibiotics, corticosteroids, immunosuppressors, or pain medications.
* Has important sensory deficits such as legally blind.
* Is currently pregnant or a nursing mother.
* Has history of, or laboratory evidence of HIV, Hepatitis B or C at Screening.
* Has laboratory evidence of Platelets < 100,000 or >600,000 k/microliter.
* Has a positive urine drug screen unless taking prescribed medication and at the discretion of the PI.
* Has a current illness that as judged by the study physician substantially increases the risks associated with performing a biopsy procedure.
* Has a history of an active bleeding disorder such as haemophilia or Von Willebrand disease.
* Is claustrophobic and/or is not eligible to perform MRI as per the MRI eligibility form.
* Has a hip or knee replacement or other medical conditions that prevents MRI research scans from being performed.
* Has a diagnosis of cognitive impairment that clearly prevents the participant from providing informed consent.
* Has a history of, or evidence of heart disease including unstable angina, myocardial infarction, congestive heart failure, cerebrovascular diseases, uncontrolled hypertension, uncontrolled cardiac arrythmias, moderate to severe valvular disease.
* Has a history or has chronic liver disease as evidenced by medical history or ALT, AST, or alkaline phosphatase twice the normal serum concentration.
* Drinks more than three drinks of alcohol per day on average.
* Has a history of, or evidence of chronic kidney disease or serum creatinine >1.1 mg/dL.

Participants must be able to speak and read English. The reason for this is for safety reasons especially as it relates to the muscle biopsy procedures. Participants will be required to provide medication history and to understand and report any problems post muscle biopsy to the research medical staff. In addition, the medical staff will be contacting the participant after the biopsies to ensure that they are recovering and do not have significant side effects for which the participant must be able to clearly verbalize for the medical staff to determine if additional observation or treatment is indicated.

Ages: 20 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled into the following age-groups: 20-29; 30-39; 40-49; 50-59; 60-69; 70-plus years with 6 participants (3 men and 3 women) in each age group.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Measure the turnover proteins in humans across tissues, age, and sex. | 21 days
  No data is available on proteins half-life that compare different tissues in humans; and this information would be important to interpret proteomic data. Comprehensively profile the turnover rates and half-lives of different proteins in human skeletal muscle.

SECONDARY OUTCOMES:
Test the hypothesis that older age is associated with diminished protein turnover. | 24 months
  Assess the turnover of proteins in muscle tissue to determine if the turnover of certain proteins and pathways are different with age.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Ferrucci, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is ongoing discussion within the NIA IRP and a plan has not been finalized yet.